CLINICAL TRIAL: NCT00502606
Title: Clinical Study :The Effect of Antibacterial Nanoparticles, Incorporated in Provisional Resin Based Cement, on S.Mutans in the Margins of Provisional Restorations
Brief Title: a Clinical Study.the Effect of Addition of Insoluble Antibacterial Nanoparticles(IABN) in Resin Base Provisional Cement
Acronym: IABN
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Ervin Weiss, Hadassah Medical Centers
Other Study IDs: 191061HMO-CTIL
Record Dates: First submitted 2007-07-16; First posted 2007-07-17 (Estimated); Last update posted 2010-01-06 (Estimated); Status verified 2009-10

CONDITIONS: Oral Rehabilitaiton; Caries; Periodontitis
Keywords: provisional restoration; antibacterial nanoparticles; cement; biofilm; bacteria; flora; plaque; dental; prosthesis
MeSH Terms: conditions — Periodontitis; Plaque, Amyloid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients with provisional crowns: the same patient would serve as control and test

SUMMARY:
The effect of Antibacterial Nanoparticles, Incorporated in cement, on S.mutans in the margins of provisional restorations is going to be examined clinically by using two kinds of provisional cement 1. cement with out antibacterial nanoparticles.

2.cement with small addition of IABN. after one week in the mouth the crowns are to be removed and examined for the presence and quantity of s. mutans. in vitro tests of the same has shown significant reduction in bacterial population around the provisional cement as compared to the regular cement.

DETAILED DESCRIPTION:
Provisional cement withholding antibacterial properties may be useful in preventing caries in the margins of provisional restorations. Covalently attached antibacterial polymers are a possible solution.

The provisional restoration is important in determine the success of the therapy. The provisional restoration protects the pulp and the dentin, and is used for diagnostic purposes. Sometimes provisional restoration can stay in the oral cavity for a long period. Through this time, the abutments must get the best biological and mechanical defense. The cement should have good mechanical properties, low solubility and good adhesion. The finishing line is a place prone to caries development due to the existence of a potential gap between the provisional restoration and the tooth.

This in vivo study will evaluate the antibacterial effect of alkylated polyethylenimine nanoparticles (IPN) incorporated to temporary cement, against S.mutans. We will compare 2 temporary cement, one with, and the other without the nano particles, using the direct technique for making provisional restoration with polymethyl methacrylate.

Baldissara et.al tested 4 kinds of temporary cements in 30 acryl resin crowns, prepared on extracted teeth. They authors found that in all 4 kinds of cements there was always a micro leakage, to some degree, in the margins of the restoration. These gap and micro leakage in restorations, contribute to restoration's failure.

Composites releasing Fluoride do not have antibacterial effect after light curing. This fact can explain why plaque tends to accumulate on composites. Polymethl metacrylate resin, the material used in direct provisional crown preparation, has a low antibacterial activity.

In the past there was an attempt to create resin composites with antibacterial activity, through incorporation of an antibacterial agent= Chlorhexidine. This agent is released from the composite, and by doing so, can cause toxicity and a decrease in the mechanical properties and in effectiveness.

Several reports have described incorporation of a methacryloyloxydodecylpyridinium bromide (MDPB) monomer in composite resins that showed no release of the incorporated monomer but still exhibited antibacterial properties.

Beith et.al tested the effect of the IPN on S.mutans. This in vitro study evaluated the antibacterial effect of alkylated polyethylenimine nanoparticles incorporated into 3 kinds of composite resins. The IPN were mixed in a low concentration of 1% w/w and cured by light polymerization. The cured samples were tested for antibacterial and mechanical properties. The addition of 1% w/w of nanoparticles did not affect significantly the flexural modulus and the flexural strength of the materials. The results indicate the IPN immobilized in resin based materials have a strong antibacterial activity on cariogenic bacteria upon contact.

The relationship between caries development and bacteria was based in the past. The disease occurs due to specific bacteria, especially from the group of mutans streptococci, ו-lactobacilli.

The assumption is that the IPN have antibacterial activity against S.mutans. Today, there is no dental material that can solve the problem of caries development in margins of provisional restorations. Many people stay with the provisional restoration for a long period in the oral cavity, in which the risk for caries development rises. Therefore there was a need to test the in vivo activity of the nanoparticles in provisional cement, on S.mutans in the margins of provisional restorations.

In the first stage of the experiment, an in vitro test using the direct contact test (DCT) will be performed. The nanoparticles will be incorporated to the cement in 3 concentrations: 0.5%, 1%, 2% , and the affect on S.mutans will be testes after 24 h, and after 14 days. The concentration will be compare to 0%. The purpose of the test is to make sure that the temporary cement with the nanoparticles supplement has an antibacterial affect against S.mutans, and that the cement without the supplement has no such activity. Furthermore, the dosages for use in vivo, will be decided based on this test.

In the next stage, an in vivo test will be performed. The temporary cement without the supplement will be placed under the provisional restoration. After a week an impression of the finishing line, And the mesial and distal walls will be taken upon a gum with sugar. The cement will be replaced with the same kind of cement, but with the IPN supplement, and will be impressed in the same manner a week later. After each appointment (2 for each patient), the gum impression will be placed on a selective S.mutans media (Mitis salivarius bacitracin,MSB( for 48h, at °37 C. Using the image-pro program, the concentration of the bacteria per area will be determined. In this way we will estimate the antibacterial activity of the supplement in the cement.

Criteria for exclusion; Appearance of allergy to the cement. Using antibiotic drug during the experiment. Mouth rinse with antibacterial properties.

The no. of participants in the experiment and the methods of analyzing the data, will be determined by a statistician after a pilot will be performed on 6 patients.

Inclusion criteria Patients who need provisional restorations.

Exclusion criteria Patients who got antibacterial therapy in the past 3 months. Patients using chlorhexidine gluconate. Pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Patients who need provisional restorations.

Exclusion Criteria:

* Patients who got antibacterial therapy in the past 3 months.
* Patients using chlorhexidine gluconate.
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: hadassah dental patients
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2007-02; Primary Completion 2010-12 (Estimated); Study Completion 2011-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Perez Davidi, DMD, Principal Investigator — Hadassah Medical Organization; Nir Sterer, DMD PhD, Study Director — Hadassah Medical Organization; Ervin Weiss, DMD, Study Chair — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization,, Jerusalem, Israel

REFERENCES:
- [Result] Beyth N, Yudovin-Farber I, Bahir R, Domb AJ, Weiss EI. Antibacterial activity of dental composites containing quaternary ammonium polyethylenimine nanoparticles against Streptococcus mutans. Biomaterials. 2006 Jul;27(21):3995-4002. doi: 10.1016/j.biomaterials.2006.03.003. Epub 2006 Mar 27. PMID 16564083
- See also: Michael Perez Davidi — http://www.mypd.co.il